CLINICAL TRIAL: NCT01363414
Title: Randomized Controlled Trial of the Effects of Sodium Hyaluronate on Wavefront Aberrations in Dry Eye Patients
Brief Title: Sodium Hyaluronate and Wavefront Aberrations in Dry Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Kaevalin Lekhanont, Department of Ophthalmology, Ramathibodi Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SVS20-THAI-05-01
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2010-09

CONDITIONS: Dry Eye
Keywords: Dry eye; Ocular aberration
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artificial tear (Experimental): One drop of preservative-free, hypotonic 0.18% sodium hyaluronate in one eye
  Interventions: Drug: 0.18% sodium hyaluronate
- Control (Placebo Comparator): one drop of sterile 0.9% sodium chloride solution in the other eye
  Interventions: Drug: 0.9% sodium chloride solution

INTERVENTIONS:
Drug: 0.18% sodium hyaluronate — one drop of preservative-free, hypotonic 0.18% sodium hyaluronate in one eye
  Other Names: Vislube®/ Vismed®
  Arms: Artificial tear
Drug: 0.9% sodium chloride solution — one drop of sterile 0.9% sodium chloride solution in the other eye
  Other Names: 0.9% NSS
  Arms: Control

SUMMARY:
Eyes with abnormal tear film function have been found to show larger optical aberrations than normal eyes which may be attributed to the unstable and irregular tear film, uneven ocular surface, and increased scatter due to the exposure of the rough surface of corneal epithelium after tear break-up.

These hypotheses have been supported by the findings that instillation of artificial tears (sodium hyaluronate preparation) in dry eye patients reduces both corneal and ocular aberrations, improving the optical quality of the retinal image.

However, the previous studies only evaluated the short-term effects of a single administration of an artificial tear but did not determine the duration of action or inflection point at which the ocular aberrations increase back to baseline. Also, there has clearly been no such clinical trial that has been a well randomized controlled study to date.

This report is the first randomized controlled trial that investigated the long-term effects of a single dose of sodium hyaluronate-based artificial tears on wavefront aberrations in patients with dry eye.

DETAILED DESCRIPTION:
Parameters used to determine treatment outcomes included ocular aberrations and severity of dry eye symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or over.
2. Documented history of bilateral dry eye for at least 3 months.
3. Schirmer's I test (without anesthesia) less than 10 mm wetting/5 minutes for each eye.
4. Tear film break-up time (TBUT) less than 10 seconds for each eye.
5. Good compliance with the study regimen and availability for the duration of the entire study period.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Contact lens wear.
3. Non-mydriatic pupil size less than 5.0 mm.
4. Other ocular surface pathologies or coexisting ocular diseases.
5. Ocular surgery or trauma within the past 4 months.
6. Use of concomitant eye drops or eye ointments within the past 2 weeks.
7. Abnormality of the nasolacrimal drainage apparatus.
8. Permanent or temporary occlusion of lacrimal puncta in any eye.
9. Known hypersensitivity to hyaluronic acid or any component used in the study.
10. Taking the following systemic medications within the previous 2 months: tricyclic antidepressive agents, anti-histaminic agents, phenothiazines, cholinergic agents, antimuscarinic agents, NSAIDs, beta-blockers, immunomodulators, anti-acneic agents, diuretics, corticosteroids and tetracyclines.
11. Very severe dry eye causing inaccurate aberrometry measurements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-01; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Ocular aberrations | 120 minutes
  A Zywave® II aberrometer which is a wavefront-sensing device based on the Hartmann-Shack principle was used to analyze monochromatic wavefront aberrations of the whole eye.

SECONDARY OUTCOMES:
Severity of dry eye symptoms | 120 minutes
  Dry eye symptoms in both eyes were graded separately by an interview based on a questionnaire inquiring about 12 symptoms: soreness, scratchiness, dryness, grittiness, burning, itchiness, ocular fatigue, lid heaviness, blurred vision, photophobia, discharge, and excess tearing, using a 0-100 mm visual analogue scale (VAS) (0 = no symptoms to 100 = severe symptoms)
Adverse reactions and complications | 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kaevalin Lekhnaont, MD, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Ramathibodi Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Lekhanont K, Chuckpaiwong V, Vongthongsri A, Sangiampornpanit T. Effects of sodium hyaluronate on wavefront aberrations in dry eye patients. Optom Vis Sci. 2014 Jan;91(1):39-46. doi: 10.1097/OPX.0000000000000101. PMID 24366433